CLINICAL TRIAL: NCT00185003
Title: Blockade of Vascular Potassium Channels During Human Endotoxemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PP02; ZONMW grant 907-00-056
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-04

CONDITIONS: Endotoxemia
Keywords: Endotoxemia; vascular potassium channels; cytokine; norepinephrine; regional blood flow,; inflammation,; ion channels,; nitric oxide synthase,; pharmacology.
MeSH Terms: conditions — Endotoxemia; Inflammation | interventions — Endotoxins; Tolbutamide; omega-N-Methylarginine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: endotoxin
Drug: Potassium channel blockers: TEA, Quinin, Tolbutamide
Drug: L-NMMA

SUMMARY:
Background: Activation of NO-synthase and vascular potassium (K) channels may play a role in the sepsis-induced attenuated sensitivity to norepinephrine. We examined whether various K channel blockers and NO-synthase inhibition could restore norepinephrine sensitivity during experimental human endotoxemia.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* drug, alcohol, nicotine abuse

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2003-01; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Hemodynamics | 24 hrs after LPS administration
Markers of Inflammation | 24 hrs after LPS administration
Cytokines | 24 hrs after LPS administration
Markers of Renal Injury | 24 hrs after LPS administration
Inducible NO synthase expression | 24 hrs after LPS administration
NO-metabolites | 24 hrs after LPS administration
Mediators of Vascular reactivity | 24 hrs after LPS administration
Sensitivity to norepinephrine | 24 hrs after LPS administration

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pickkers, MD, PhD, Principal Investigator — Radboud University Medical Center

REFERENCES:
- [Result] Pickkers P, Dorresteijn MJ, Bouw MP, van der Hoeven JG, Smits P. In vivo evidence for nitric oxide-mediated calcium-activated potassium-channel activation during human endotoxemia. Circulation. 2006 Aug 1;114(5):414-21. doi: 10.1161/CIRCULATIONAHA.105.590232. Epub 2006 Jul 24. PMID 16864730